CLINICAL TRIAL: NCT00924313
Title: A Pilot Study of 11C-Acetate Positron Emission Tomography (PET) and 3 Telsa Magnetic Resonance Imaging (MRI) in Men With Prostate Cancer Undergoing Prostatectomy
Brief Title: Positron Emission Tomography and Magnetic Resonance Imaging for Prostate Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Peter Choyke, M.D., Principal Investigator, National Institutes of Health Clinical Center (CC)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 080226; 08-C-0226; NCT00771550 (obsolete NCT alias)
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Results first posted 2012-08-17 (Estimated); Last update posted 2017-07-11 (Actual); Status verified 2017-06

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; C-11 Acetate; PET
MeSH Terms: conditions — Prostatic Neoplasms | interventions — carbon-11 acetate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 11C-acetate for Prostate Cancer Patients (Experimental): 11C-acetate positron emission tomography (PET)/computed tomography (CT)for 30 minutes, intravenous bolus injection
  Interventions: Drug: (C-11 Acetate)

INTERVENTIONS:
Drug: (C-11 Acetate) — 11C-acetate positron emission tomography (PET)/computed tomography (CT)for 30 minutes, intravenous bolus injection

SUMMARY:
Background:

* Prostate cancers are difficult to see on most imaging studies such as X-rays, computed tomography (CT) scans, conventional magnetic resonance imaging (MRI) scans and conventional positron emission tomography (PET) scans.
* An experimental radioactive tracer called 11C-acetate accumulates in prostate tumor cells and may help find prostate cancers more accurately than other imaging methods.

Objectives:

* To determine the accuracy of prostate tumor imaging using the tracer 11C-acetate.

Eligibility:

* Patients 18 years of age and older who are undergoing surgery for localized prostate cancer at the National Institutes of Health (NIH) Clinical Center.

Design:

* Patients have a positron emission tomography (PET scan). For this test, an intravenous (IV) line is placed in the patient's arm and the patient lies on a table inside the donut shaped scanner. (11)C-acetate is injected into the vein through the catheter and images of the lower pelvis and abdomen are obtained over 30 minutes.
* Patients have an endorectal coil MRI scan. For this test, a tube is placed in the rectum, just behind the prostate, to increase the amount of signal received by the magnetic resonance (MR) unit. Other coils may be wrapped around the pelvis to further improve the quality of the scan. The patient lies on the scanning table for about 75 to 90 minutes while images are obtained. During the scan, a contrast agent called gadolinium is injected through an intravenous (IV) line to brighten the images.

DETAILED DESCRIPTION:
Background:

* Accurate localization of prostate cancer (PC) is important in developing targeted minimally invasive therapies. While T2 weighted imaging, dynamic contrast enhanced (DCE) imaging, diffusion weighted imaging (DWI), and magnetic resonance (MR) spectroscopy imaging performed at 3T is a useful technique for localizing prostate cancer, it has limitations both in sensitivity and specificity.
* Positron emission tomography (PET) radiopharmaceuticals are more sensitive than magnetic resonance imaging (MRI) for the detection of cancers; however, the resolution of PET is inferior to MRI. Therefore, a combined PET/MR approach might be desirable.
* We propose to evaluate the utility of a PET radiopharmaceutical, (11C) acetate ((11C)AC) for the detection of PC within the prostate and compare its distribution with T2 weighted imaging, dynamic contrast enhanced (DCE) imaging, diffusion weighted imaging (DWI), and MR spectroscopy imaging preformed at 3T.
* Unlike fludeoxyglucose F18(18F)FDG, a routinely used PET radiopharmaceutical which is excreted by the urinary system and accumulates in the bladder, limiting its utility in pelvic imaging, (11C)AC has low physiologic distribution in the pelvis. Several studies involving small numbers of patients have demonstrated that (11C)AC PET imaging can localize in pelvic nodes involved with prostate cancer (PC).
* Dynamic (11C)AC PET/CT examination will be performed in patients with biopsy proven prostate cancer (estimated enrollment 40) who will also undergo prostate/pelvic 3T endorectal coil MR/magnetic resonance spectroscopic imaging (MRSI) followed by surgical resection (+/- pelvic lymphadenectomy).
* Histological comparison with the PET/CT and MRI results will be conducted. This study of (11C)AC in PC will permit the direct comparison of MR/MRSI and (11C)AC PET/CT in the detection of prostate cancer within the prostate.

Objectives:

Primary Objective:

- To compare the biodistribution of (11C) acetate ((11C)AC) PET/CT imaging in tumor and non-tumorous regions of the prostate in patients with known prostate cancer.

Secondary Objective:

* To examine the diagnostic accuracy of the standardized uptake value (SUV) of (11C)AC obtained using PET/CT imaging for detecting region (sextant)-specific malignancy using receiver operating curves (ROC).
* To examine whether pelvic biodistribution of (11C)AC PET/CT imaging predicts sextant-specific malignancy better than T2 weighted imaging, dynamic contrast enhanced (DCE) imaging, diffusion weighted imaging (DWI), and MR spectroscopy (MRS) imaging performed at 3T.
* To evaluate for potential physiological effects of (11C)AC
* To correlate the intensity of (11C)AC uptake with histopathologic Gleason Grade
* Tabulate the incidence of extraprostatic lesions accumulating(11C)AC PET/CT detection which are suspicious for extraprostatic disease by comparing suspicious lesions on (11C)AC PET/CT with standard of care diagnostic imaging modalities, additional biopsy results, or clinical follow-up performed at the discretion of the referring physician.

Eligibility:

* Participants must be scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the National Institutes of Health (NIH) Clinical Center.
* Recent (within 12 months of study entry) biopsy indicating the presence of adenocarcinoma of the prostate gland
* Participant must be 18 years or older
* Serum creatinine within 1 week prior to MR imaging less than or equal to 1.8mg/dl AND epidermal growth factor receptor (eGFR) must be greater than 30 ml/min/1.73m^2
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 or 1
* Participants may not have received androgen deprivation therapy or pelvic radiation therapy

Design:

* Participants with prostate cancer scheduled for prostatectomy at the NIH Clinical Center will undergo 30-minute dynamic (11C)AC PET/CT imaging, and endorectal coil/pelvic T2 weighted, DCE, DWI, and MRS imaging performed at 3T.
* We will accrue 40 participants to this study.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participant must be scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the National Institutes of Health (NIH) Clinical Center.
* Recent (within 12 months of study entry) trans-rectal biopsy indicating the presence of adenocarcinoma of the prostate gland in which at least sextant biopsies were obtained. Knowledge of the location of each specimen is required for inclusion.
* Participant must be 18 years or older.
* Serum creatinine within 1 week prior to magnetic resonance (MR) imaging less than or equal to 1.8mg/dl AND epidermal growth factor receptor (eGFR) must be greater than 30 ml/min/1.73 m^2
* Eastern Cooperative Oncology Group (ECOG) Performance score of 0 or 1.
* Ability to provide informed consent. All patients must sign a document of informed consent indicating their understanding of the investigational nature and risks of the study before any protocol related studies are performed.

EXCLUSION CRITERIA:

* Known allergy to gadolinium or acetate.
* Participants for whom participating would significantly delay the scheduled standard of care therapy.
* Participants with any coexisting medical or psychiatric condition that is likely to interfere with study procedures and/or results are excluded.
* Participants with severe claustrophobia.
* Patients with contraindications to magnetic resonance imaging (MRI)
* Patients weighing greater than 136 kg (weight limit for scanner table).
* Patients with pacemakers, cerebral aneurysm clips, shrapnel injury, or other implanted electronic devices or metal not compatible with MRI.
* Patients with contraindication to endorectal coil placement
* Severe hemorrhoids.
* Surgically absent rectum.
* Other medical conditions deemed by the principal investigator (PI) or associates to make the patient ineligible for protocol procedures.
* Patients who have previously received radiation therapy to the pelvis.
* Patients who have received androgen deprivation therapy.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — * Participant must be scheduled to undergo standard of care prostatectomy for presumed localized prostate cancer at the National Institutes of Health (NIH) Clinical Center.
  * Recent (within 12 months of study entry) trans-rectal biopsy indicating the presence of adenocarcinoma of the prostate gland in which at least sextant biopsies were obtained. Knowledge of the location of each specimen is required for inclusion.
Enrollment: 40 (Actual)
Dates: Start 2008-09-10 (Actual); Primary Completion 2011-04-19 (Actual); Study Completion 2011-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Choyke, M.D., Principal Investigator — National Cancer Institute, National Institutes of Health
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Oyama N, Miller TR, Dehdashti F, Siegel BA, Fischer KC, Michalski JM, Kibel AS, Andriole GL, Picus J, Welch MJ. 11C-acetate PET imaging of prostate cancer: detection of recurrent disease at PSA relapse. J Nucl Med. 2003 Apr;44(4):549-55. PMID 12679398
- [Background] Jung JA, Coakley FV, Vigneron DB, Swanson MG, Qayyum A, Weinberg V, Jones KD, Carroll PR, Kurhanewicz J. Prostate depiction at endorectal MR spectroscopic imaging: investigation of a standardized evaluation system. Radiology. 2004 Dec;233(3):701-8. doi: 10.1148/radiol.2333030672. PMID 15564406
- [Result] Mena E, Turkbey B, Mani H, Adler S, Valera VA, Bernardo M, Shah V, Pohida T, McKinney Y, Kwarteng G, Daar D, Lindenberg ML, Eclarinal P, Wade R, Linehan WM, Merino MJ, Pinto PA, Choyke PL, Kurdziel KA. 11C-Acetate PET/CT in localized prostate cancer: a study with MRI and histopathologic correlation. J Nucl Med. 2012 Apr;53(4):538-45. doi: 10.2967/jnumed.111.096032. Epub 2012 Feb 17. PMID 22343504

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 11C-acetate for Prostate Cancer Patients
Started | 40
Completed | 39
Not Completed | 1
Not completed — not imaged due to failed tracer imaging | 1

BASELINE CHARACTERISTICS:
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 33
  >=65 years | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.97 (6.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 36
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 28
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Number; unit: participants]
  United States | 40
Interval Between Magnetic Resonance Imaging and Prostatectomy [Mean (Full Range); unit: Days] — Prostatectomy is a partial or total removal of the prostate gland. Population: One patient was not imaged due to failed tracer synthesis. One patient was not evaluable due to inadequate registration between the transmission scan and magnetic resonance imaging.
  Days
    number analyzed (Participants) | 38
    (all) | 54 [2 to 155]
Days to Radical Prostatectomy [Mean (Full Range); unit: Days] — Radical prostatectomy is removal of the entire prostate gland. and additional tissue Population: One patient was not imaged due to failed tracer synthesis. One patient was not evaluable due to inadequate registration between the transmission scan and magnetic resonance imaging.
  Days
    number analyzed (Participants) | 38
    (all) | 10.5 [1 to 34]

OUTCOME MEASURES:

1. Primary Outcome: Compare the Biodistribution of 11C-acetate Positron Emission Tomography (PET)/Computed Tomography (CT) Imaging in Tumor and Non Tumorous Regions of the Prostate
Description: Standard uptake values (SUV) measurements of 11C-acetate will be obtained in each sextant (e.g. region) on each patient. Sextant-specific malignancy will be determined pathologically based on a subsequent prostatectomy. Initially, on each patient, we will, average SUV measurements in tumor and non-tumor regions (i.e., sextants with malignancy and no malignancy, respectively). The patient average SUV measurements across tumors and non-tumor regions will then be compared using a paired t-test.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 39
ng/mL
  Tumor region | 4.4 (2.05)
  Non-tumorous region | 2.1 (0.94)

2. Secondary Outcome: Count of Participants With Adverse Events
Description: Here is the number of participants with adverse events. For the detailed list of adverse events see the adverse event module.
Time Frame: 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 39
Participants | 14

3. Secondary Outcome: Diagnostic Accuracy of the Standardized Uptake Value of [11C]AC Obtained Using Positron Emission Tomography (PET)/Computed Tomography (CT) for Detecting Region (Sextant)-Specific Malignancy Using Receiver Operating Curves (ROC) for a Lesion >0.9cm
Description: The diagnostic accuracy of 11C-Acetate PET/CT imaging in prostate cancer was compared with multi-parametric magnetic resonance imaging (MP-MRI) using sector based analysis, generating receiver-operating-characteristic (ROC) curves (plots of 1-specificity versus sensitivity) for both modalities.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Number (95% Confidence Interval); unit: Percentage ROC curve
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
Percentage ROC curve
  PET sensitivity | 62 [59 to 65]
  MRI sensitivity | 82.3 [79 to 85]
  PET specificity | 80 [78 to 82]
  MRI specificity | 95 [92 to 97]

4. Secondary Outcome: Pelvic Biodistribution of [11C]AC Positron Emission Tomography (PET)/Computed Tomography (CT) Imaging
Description: Pelvic biodistribution was obtained for the prostate tumor, normal prostate and benign prostatic hyperplasia (BPH). Uptake is expressed in standardized uptake value (SUV).
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
SUV
  Prostate tumor | 4.4 (2.05)
  Normal tumor | 2.1 (0.943)
  Benign prostatic hyperplasia (BPH) | 4.8 (2.01)
Statistical Analysis 1: Comparison: 11C-acetate for Prostate Cancer Patients; Test type: Superiority; p < 0.0001, Spearman rank correlation — The reported p-value is representative of the difference in levels of the histopathologic confirmed tumor and normal prostate tissue
Statistical Analysis 2: Comparison: 11C-acetate for Prostate Cancer Patients; Test type: Superiority; p = 0.65, Spearman rank correlation — The reported p-value is representative of the BPH high uptake level

5. Secondary Outcome: Count of Participants With Physiological Effects of [11C]AC
Description: Buildup of positron emission tomography (PET) radiopharmaceuticals excreted by the urinary system can accumulate in the bladder and limit pelvic imaging. This effect contributes to low physiologic distribution in the pelvis.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
Participants | 1

6. Secondary Outcome: Incidence of Extraprostatic Lesions Accumulating [11C]AC Positron Emission Tomography (PET)/Computed Tomography (CT) Detection
Description: Suspicious lesions noted on biopsy were compared with standard care imaging diagnostic modalities, additional biopsies, and/or clinical follow up performed at the discretion of the referring physician.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Count of Participants; unit: Participants
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
Participants | 1

7. Secondary Outcome: Standardized Uptake Value (SUV) of Grouping Tumors Based on Gleason Score
Description: Intensity [11C]AC uptake with histopathologic Gleason grade were done with a Spearman rank correlation following prostatectomy. Two biopsies were performed and graded according to tumor pattern. The two grades were added together for a final Gleason score. Gleason score equal to or less than 3+4 is considered low risk. Gleason score equal to or greater than 4+3 is considered high-risk.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Mean (Standard Deviation); unit: SUV
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
SUV
  Gleason scores 3+4 and below | 4.2 (1.8)
  Gleason scores 4+3 and above | 4.9 (3.1)
Statistical Analysis 1: Comparison: 11C-acetate for Prostate Cancer Patients; Test type: Superiority; p = 0.55, Spearman rank correlation

8. Secondary Outcome: Lesion Based Sensitivity Analysis Using Positron Emission Tomography (PET)/Computed Tomography (CT), Multi-parametric Magnetic Resonance Imaging (MP-MRI), Diffusion Weighted-Magnetic Resonance Imaging (DW-MRI), and DCE-MRI.
Description: PET/CT, MP-MRI, DW-MRI, and dynamic contrast enhanced magnetic resonance imaging (DCE-MRI) were used to detect lesion sensitivity.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Number (95% Confidence Interval); unit: percentage of sensitivity
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
percentage of sensitivity
  PET/CT | 73.4 [70 to 75]
  MP-MRI | 88.5 [82 to 92]
  DW-MRI | 80 [76 to 85]
  DCE-MRI | 55 [50 to 61]

9. Secondary Outcome: 11C-Acetate Standardized Uptake Value (SUV)Max and Serum Prostate Specific Antigen (PSA) Levels Using Spearman Correlation
Description: Tumor foci was histopathologically identified and tested to determine SUVmax relative to PSA levels. PSA normal range is 0-4ng/mL.
Time Frame: 2 years
Population: One patient was not imaged because of failed tracer synthesis.
Measure: Mean (Standard Deviation); unit: SUVmax
Arm/Group | 11C-acetate for Prostate Cancer Patients
Number analyzed (Participants) | 38
SUVmax
  PSA level <4 ng/ml | 3.7 (2.0)
  PSA level 4-10 ng/ml | 4.9 (2.3)
  PSA level >10ng/ml | 5.1 (0.8)
Statistical Analysis 1: Comparison: 11C-acetate for Prostate Cancer Patients; Test type: Superiority; p = 0.407, Spearman rank correlation

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 11C-acetate for Prostate Cancer Patients
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 14/40
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 11C-acetate for Prostate Cancer Patients (N=40)
Constitutional Symptoms-Other (Specify, Funny smell) (General disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 10 (10)
Vomiting (Gastrointestinal disorders) | 1 (1)
Syncope (fainting) (Nervous system disorders) | 1 (1)
Pain: Back (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain: Extremity-limb (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No